CLINICAL TRIAL: NCT06371833
Title: A Multicentric Study Evaluating Clinical and Radiological Outcomes of PRIMA Humeral Stem in Total Shoulder Arthroplasty
Brief Title: PRIMA EU Retrospective & Prospective
Status: Recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: S-52
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Arthroplasty; Replacement; Shoulder
Keywords: TSA; RSA; Shoulder replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients requiring a primary TSA or RSA: Device: PRIMA humeral stem in anatomic or reverse configuration Shoulder arthroplasty according to the instruction for use.
  Interventions: Device: Shoulder Arthroplasy with PRIMA humeral stem

INTERVENTIONS:
Device: Shoulder Arthroplasy with PRIMA humeral stem — Data collection of population that underwent a total shoulder arthroplasty with PRIMA humeral stem (anatomic configuration or reverse configuration)

SUMMARY:
This clinical study aims at evaluating clinical, radiographic and patient-reported outcomes after total anatomic or reverse shoulder replacement using PRIMA humeral stem up to 24 months after surgery, in order to assess the short-term performance of the implant. Furthermore, the objective is also to collect short-term data on the survivorship of the implant and the incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Full skeletal maturity;
3. Life expectancy over 24 months;
4. Patient's joint anatomically and structurally suited to receive the selected implants and functional deltoid muscle;
5. Patient meets at least one of the following indications:

   For Anatomic configuration:
   * non-inflammatory degenerative joint disease (i.e., osteoarthritis);
   * inflammatory arthritis of the glenohumeral joint including rheumatoid arthritis;
   * avascular necrosis of the humeral head;
   * cuff tear arthropathy (CTA Heads only);

   For Reverse configuration:
   * rotator cuff tear arthropathy;
   * osteoarthritiswith rotator cuff tear;
   * rheumatoid arthritis with rotator cuff tear;
   * massive irreparable rotator cuff tear;
6. Patient is able to understand the conditions of the study, to comply with the prescribed rehabilitation as well as willing to perform all scheduled follow-up visits;
7. Patient has signed the Informed Consent form previously approved by the Ethics Committee before study activities.

Exclusion Criteria:

1. Patients who lack capacity to be able to provide informed consent to participate in the study.
2. Local or systemic general infection;
3. Septicaemia;
4. Persistent acute or chronic local or systemic osteomyelitis;
5. Confirmed neurologic lesion compromising shoulder joint function;
6. Deltoid muscle insufficiency;
7. Poor meta-epiphyseal bone stock compromising stability of the implant (severe fracture of the proximal humerus, meta-epiphyseal pseudoarthrosis, osteoporosis, osteomalacia, extended bone loss after previous prosthetic or non-prosthetic surgery);
8. Affected by malignant cancer with life expectancy less than 2 years or where cancer treatment might affect the normal postoperative course;
9. Serious muscular, neurological, or arterial vascular diseases compromising stability of the implant;
10. Proximal humerus fracture sequelae with inadequate bone stock;
11. Vascular or nerve diseases affecting the concerned limb;
12. Metabolic disorders which may impair fixation and stability of the implant;
13. Any concomitant disease that might affect the implanted prosthesis;
14. Metal hypersensitivity to implant materials (CoCrMo);
15. Patient with significant renal impairment;
16. Lower mobility issues that may affect the study evaluation;
17. Unwillingness or inability (due to physical or mental issues) to comply with rehabilitation and to return for follow-up visits and any psychiatric illness that would prevent comprehension of the details and nature of the study;
18. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant;
19. Any clinically significant pathology based on the medical history that the Investigator feels may affect the study evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible study population consists of 60 adult patients requiring a primary Total Shoulder Arthroplasty (TSA) or Reverse Shoulder Arthroplasty (RSA).
  The decision to use PRIMA humeral stem has been taken by the Investigator prior to, and independently from, the decision to include the subject in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Costant Murley Score (CS) | From preoperative (baseline) to 24-month follow-up.
  The primary endpoint is to assess the change of Constant Murley Score (CS). Constant score (CS) is a clinical method of shoulder functional assessment that allows individual-parameter assessments to be combined with an overall 100-point scoring system. The final result is graded, with the normalized 100-point shoulder score, as excellent (85 to 100 points), good (71 to 84 points), fair (56-70), poor (0-55). The weighted Constant score is calculated as a percentage of norm

SECONDARY OUTCOMES:
Changes in the American Shoudler and Elbow Surgeons (ASES) score | From preoperative (baseline) to 24-month follow-up.
  American Shoulder and Elbow Surgeons (ASES) score contains a patient self-report section and a section used by medical professionals to record physical examination findings to assess patients with shoulder pathologies. It is a patient self-evaluation questionnaire that takes approximately 5 minutes to complete and consists of 2 dimensions: pain and activities of daily living. The pain score is calculated from the single pain question and the function score from the sum of the 10 questions addressing function. The pain score and function composite score are weighted equally (50 points each) and combined for a total score out of a possible 100 points [with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition].
Changes in Range of Motion measures | From preoperative (baseline) to 24-month follow-up.
  Range of active movements and passive movements, where available, are recorded for:
  * Forward elevation (passive and active);
  * External rotation with arm at the side (passive and active);
  * External rotation in 90° of abduction (passive and active);
  * Internal rotation (passive and active).
Radiographic stability of the humeral component | From immediate postoperative (baseline) to 24-months follow-up
  All radiographs performed during the clinical study fall within site's standard of care. Views collected may include antero-posterior (AP) and axillary or scapula y view. In case CT scans, sonography, MRI are performed at specific time-points, they can be made available for collection and evaluation.
  Imaging are collected to evaluate the radiographic performance of the device.
Survival rate (Kaplan-Meier estimate) | From immediate post-operative to 24-months follow-up.
  The Kaplan-Meier method is used to estimate the survivorship of the implant. Here, point estimates, 95% confidence bands and survival curve are provided.
  In case PRIMA humeral stem is revised for any reason, the patient will be followed up to the last follow up to evaluate the survival of the remaining component.
Incidence, type and severity of Adverse Events and Adverse Device Effects | From surgery to 24-months follow-up.
  Incidence, type and severity of all the Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) occurred at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Castagna, Principal Investigator — Humanitas Rozzano, Italy; Paolo Paladini, Principal Investigator — Unit of Shoulder Surgery Romagna/ Cervesi Hospital, Italy; Jörn Kircher, Principal Investigator — ATOS Klinik Fleetinsel Hamburg, Germany; Amar Malhas, Principal Investigator — Royal Berkshire NHS Trust, UK; Fernando Marco Martinez, Principal Investigator — Hospital Clinico San Carlos, Spain; Iain Packham, Principal Investigator — North Bristol NHS Trust, UK
Locations (1):
- Unit of Shoulder Surgery Romagna/ Cervesi Hospital, Italy, Cattolica, Rimini, Italy